CLINICAL TRIAL: NCT04319692
Title: Effect of Fermented Prunus Mume Vinegar on Improvement of Fatigue: a Randomized Controlled Trial
Brief Title: Effect of Fermented Prunus Mume Vinegar on Improvement of Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-2018-030
Record Dates: First submitted 2020-03-21; First posted 2020-03-24 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fermented Prunus Mume Vinegar group (Experimental): This group takes Fermented Prunus Mume Vinegar for 8 weeks.
  Interventions: Dietary Supplement: Fermented Prunus Mume Vinegar group
- Placebo group (Placebo Comparator): This group takes placebo for 8 weeks.
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Fermented Prunus Mume Vinegar group — This group takes Fermented Prunus Mume Vinegar for 8 weeks
  Arms: Fermented Prunus Mume Vinegar group
Dietary Supplement: Placebo group — This group takes placebo for 8 weeks.
  Arms: Placebo group

SUMMARY:
The investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of Fermented Prunus Mume Vinega on Improvement of Fatigue in adults for 8 weeks.

DETAILED DESCRIPTION:
Previous studies have indicated that Fermented Prunus Mume Vinega may have the ability to improve fatigue. Therefore, the investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of tFermented Prunus Mume Vinega on Improvement of Fatigue in adults; the safety of the compound are also evaluate. The Investigators examine fatigue severity scale, lactate, creatinine kinase, urinary malondialdehyde at baseline, as well as after 4 and 8 weeks of intervention. Sixty adults were administered either 600 mg of Fermented Prunus Mume Vinega or a placebo each day for 8 weeks;

ELIGIBILITY:
Inclusion Criteria:

* Those who complain of fatigue for more than 1 month
* Fatigue Severity Scale 3 points or more

Exclusion Criteria:

* chronic hepatitis B or C infection
* being treated for hypothyroidism or hyperthyroidism
* more than twice the normal upper limit of Creatinine
* Liver enzyme value is more than twice the normal upper limit
* Uncontrolled diabetes (over 160 mg / dl of fasting blood sugar)
* Uncontrolled hypertension (more than 160/100 mmHg, measured after 10 minutes of stability in subjects) or those with heart disease, such as angina or myocardial infarction
* taking medications that affect fatigue within the past 1 month (psychiatric drugs such as Chinese medicine, soy drugs, depression, beta-blockers, steroids, hormones, etc.). However, intermittent medication due to sleep disorders is excluded.
* a history of gastrointestinal resection or complain of severe gastrointestinal symptoms such as heartburn and indigestion
* already have participated in or plan to participate in another drug clinical trial
* Alcohol abusers
* pregnant, lactating or have a pregnancy plan during the clinical trial period
* allergic reactions to Fermented Prunus Mume Vinegar
* A person deemed inappropriate by the researcher for other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-03-19 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Fatigue severity scale | 8 weeks
  Fatigue severity scale, minimum~maximum values (1~7), higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Lactate level | 8 weeks
  Lactate level (mg/dL)
Creatinine kinase level | 8 weeks
  Creatinine kinase level (IU/L)
Urinary malondialdehyde level | 8 weeks
  Urinary malondialdehyde level (mmol/mg Cr)

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeungsangnam-do, South Korea

REFERENCES:
- [Derived] Choi JI, Lee YL, Lee SY. Efficacy and safety of fermented Prunus mume vinegar on fatigue improvement in adults with unexplained fatigue: A randomized controlled trial. Front Nutr. 2022 Nov 9;9:990418. doi: 10.3389/fnut.2022.990418. eCollection 2022. PMID 36438753